CLINICAL TRIAL: NCT04877964
Title: Ultrasound Measured Epidural Depth for Midline Approach in Pediatric Patients With Scoliosis: Prospective Observational Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2021-0266
Record Dates: First submitted 2021-04-29; First posted 2021-05-07 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pediatric patients with scoliosis: Patients aged 3-14 years with scoliosis and who request epidural analgesia
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Using ultrasound with transverse median and paramedian sagittal oblique approach, the screens that show the target epidural space in the center are obtained and stored for evaluation.

SUMMARY:
The purpose of this study was to

1. investigate the degree of agreement between the ultrasound-measured depth (in the transverse median and paramedian sagittal oblique plane) and the actual depth to the epidural space in pediatric patients with scoliosis.
2. investigate the quality of ultrasound view for detecting ligamentum flavum and dura mater.

ELIGIBILITY:
Inclusion Criteria:

1. pediatric patients (aged 3-14 years) with scoliosis (cobb angle >10 degree) scheduled for correctional osteotomy of the lower extremity and requesting epidural analgesia for postoperative pain control

Exclusion Criteria:

1. Contraindications to epidural analgesia (local infection, blood clotting disorder, anatomical abnormality, sepsis, etc.)
2. If all of the parents of the subject are foreigners or illiterate (if the parents of the subject can not read the agreement)

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients (aged 3-14 years) with scoliosis (cobb angle >10 degree) scheduled for correctional osteotomy of the lower extremity and requesting epidural analgesia for postoperative pain control
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2021-06-08 (Estimated); Primary Completion 2023-06-08 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
the degree of agreement between the ultrasound-measured depth and the actual depth to the epidural space | Ultrasound image, which is obtained before epidural Touhy needle insertion, will be evaluated within 1 week after epidural Touhy needle insertion
  the degree of agreement between the ultrasound-measured depth (in the transverse median and paramedian sagittal oblique plane) and the actual depth to the epidural space in pediatric patients with scoliosis.
the quality of ultrasound view for detecting ligamentum flavum and dura mater (in the transverse median and paramedian sagittal oblique plane) | Ultrasound image, which is obtained before epidural Touhy needle insertion, will be evaluated within 1 week after epidural Touhy needle insertion
  the quality of ultrasound view for detecting ligamentum flavum and dura mater (in the transverse median and paramedian sagittal oblique plane).
  Good: The distinction is clear and visible Fair: Visible by adjusting the probe Poor: Observation is difficult even when the probe is adjusted

CONTACTS AND LOCATIONS:
Overall Officials: Hye Jin Kim, MD, Principal Investigator — Department of Anesthesiology and Pain Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Choi YS, Jang J, Kim HY, Lee B, Kim EJ, Yoon HJ, Lee J, Kim HJ. Ultrasound estimates of the epidural depth in the paramedian sagittal oblique and transverse median planes: the correlation between estimated and actual depth to the epidural space in children with scoliosis. Reg Anesth Pain Med. 2024 Dec 2;49(12):883-888. doi: 10.1136/rapm-2023-105149. PMID 38160017